CLINICAL TRIAL: NCT06339567
Title: Evaluation of the Venous Thrombotic Biological Profile of Different PCOS Phenotypes: French Cross-sectional Study
Acronym: Hemo-PCOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 671_Hemo-PCOS
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thrombotic profil (Other)
  Interventions: Diagnostic Test: Thrombotic profile

INTERVENTIONS:
Diagnostic Test: Thrombotic profile — several thrombotic biological marker will be dosed in blood. (C protein, S protein, CRP us, Factor VIII, TFPI , nAPCsr, SHBG, nTMsr)

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder of women of childbearing age. PCOS can be individualized into several phenotypes, taking into account in particular the presence of hyperandrogenism, insulin resistance and BMI. Hyperandrogenism and insulin resistance appear to be important factors in the development of cardiovascular cardiovascular disease. In addition, patients frequently use anti-androgenic and/or contraceptive treatments contraceptives, such as combined hormonal contraception (CHC), the use of which is associated with an increased cardiovascular and thrombo and venous thrombosis (VTE). A meta-analysis published in 2020 by Gariani et al.

based on three large studies, estimated the risk of VTE in women with PCOS after adjustment for obesity and hormone therapy. This risk was significantly higher compared with women without PCOS (pooled OR 1.89, CI95% 1.60-2.24). No study has looked specifically investigated the risk of VTE according to different PCOS phenotypes. Such data would be very useful in clinical practice, as it would enable monitoring, contraceptive treatment and anti-androgenic anti-androgen treatment according to the PCOS phenotype, while limiting risks. Assessing the differences PCOS phenotypes is limited by the large sample size required. required. VTE is a rare event in women of childbearing age, and the number of PCOS phenotypes is high.

PCOS phenotypes. Intermediate markers of VTE risk are used in these situations. These markers are thrombin generation tests (notably ETP) and their sensitivity to activated protein C (nAPCsr) and thrombomodulin (nTMsr), as well as sex-hormone binding globulin (SHBG).

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 35 years of age at the time of inclusion;
* Able to give non-opposition
* Strong suspicion of PCOS according to 2023 recommendations
* Have stopped hormonal contraception for at least 3 months or insulin-sensitizing treatment for at least 3 months.
* Fasting for at least 12 hours.
* Be affiliated to a health insurance scheme.
* French-speaking

Exclusion Criteria:

* Already included in a type 1 interventional research protocol (RIPH1).
* Be under guardianship or curatorship
* Deprived of liberty
* Under court protection
* Pregnant (positive urine or blood pregnancy test), or within 3 months of post-partum or post abortum, or breastfeeding (or within 3 months of weaning)
* Using hormonal contraception or insulin-sensitizing therapy (a wash-out of at least 3 months before inclusion).
* Have a personal history of VTE or known thrombophilia.
* Current anticoagulant or antiaggregant treatment or treatment stopped less than one month before inclusion.
* Have a severe personal medical history in the previous 6 weeks (fracture, infection, hospitalization, surgery, cardiovascular event, cancer).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2029-02-07 (Estimated)

PRIMARY OUTCOMES:
biological procoagulant profile | one year
  Evaluation of the biological procoagulant profile in women of childbearing age with PCOS, in relation to the presence or absence of insulin resistance, by comparing FTE levels between women with PCOS and women without PCOS. the presence or absence of insulin resistance, by comparing ETP levels between women with PCOS without and with insulin resistance

SECONDARY OUTCOMES:
Insuline resistance and weight | 1 year
  Estimate the prevalence of overweight, obesity, and insulin resistance in women with with PCOS
comparison of procoagulant profile depending on insulin resistance | 1 year
  comparison of procoagulant biomarker for women with or without insulin resistance
comparison of procoagulant profile depending on hyperangrogenism | 1 year
  comparison of procoagulant biomarker for women with or without hyperangrogenism
comparison of procoagulant profile depending on PCOS phenotype | 1 year
  comparison of procoagulant biomarker depending on PCOS phenotype
comparison of procoagulant profile depending on AMH Rate | 1 year
  comparison of procoagulant biomarker depending on AMH Rate
comparison of QoL score depending on PCOS phenotype | 1 year
  comparison of PCOS-QoL, SF36 and HADS scores depending on PCOS phenotype

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France, France

IPD SHARING:
Plan to Share IPD: No